CLINICAL TRIAL: NCT04786366
Title: Natural History and Patient Journey in Atrial Fibrillation: a Nationwide Linked Electronic Health Records Study of 5.6 Million Individuals.
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University College, London (Other)
Responsible Party: Sponsor
Other Study IDs: ISAC17_205
Record Dates: First submitted 2020-12-04; First posted 2021-03-08 (Actual); Last update posted 2021-03-08 (Actual); Status verified 2021-03

CONDITIONS: Atrial Fibrillation; Epidemiology
Keywords: Atrial Fibrillation; healthcare contacts; Electronic Health Records; epidemiology; comorbidity; health inequality
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: The study does not have an intervention, but observe the AF incidence of the UK disease-free population — The study does not have an intervention, but observe the AF incidence of the UK disease-free population.

SUMMARY:
The trajectory of atrial fibrillation (AF) patients within the national health system and their recent temporal trends remains to be fully elucidated. To study the AF incidence, mortality and case-fatality, the investigators implemented a longitudinal cohort study with the linked electronic health records of 5.6 million population in the UK from 1998 to 2016 (CALIBER). A matched case-control study design was used to investigate the causes of hospitalization and death comparing individuals with and without incident AF.

ELIGIBILITY:
Inclusion Criteria:

* The investigators identify individuals aged 18 years or older and registered in the current primary care practice for at least one year.

Exclusion Criteria:

* Individuals are excluded if they had a prior history of AF before study entry.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The investigators implement two study designs, first a longitudinal cohort study to assess AF incidence and second a matched case-control study for mortality, cause of death and hospitalization.
  The investigators identify individuals aged 18 years or older and registered in the current primary care practice for at least one year. Individuals are excluded if they had a prior history of AF before study entry. For the nested case-control study, controls are matched to incident AF patients according to sex and age (10-year age strata).
Sampling Method: Non-Probability Sample
Enrollment: 5601803 (Actual)
Dates: Start 1998-01-01 (Actual); Primary Completion 2016-05-31 (Actual); Study Completion 2021-06-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of Atrial fibrillation | Jan 1st 1998 - May 31st 2016
  AF incidence in the population
Mortality of Atrial fibrillation | Jan 1st 1998 - May 31st 2016
  Mortality among AF patients

REFERENCES:
- [Derived] Chung SC, Schmit AF, Lip GYH, Providencia R. Electronic health record-wide association study for atrial fibrillation in a British cohort. Front Cardiovasc Med. 2023 Sep 28;10:1204892. doi: 10.3389/fcvm.2023.1204892. eCollection 2023. PMID 37840952